CLINICAL TRIAL: NCT04554225
Title: Pulmonary Disease Requiring Ambulatory Oxygen Therapy -Resilience and Quality of Life
Acronym: koti-happi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 507A023
Record Dates: First submitted 2020-08-26; First posted 2020-09-18 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Disease
Keywords: resilience; psychological; quality of life; oxygen inhalation therapy; lung diseases
MeSH Terms: conditions — Lung Diseases | interventions — nitrox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary disease patients: Patients with COPD or other pulmonary disease starting to use ambulatory oxygen therapy
  Interventions: Drug: Oxygen gas

INTERVENTIONS:
Drug: Oxygen gas — Oxygen administered to a patient using ambulatory oxygen
  Other Names: ambulatory oxygen

SUMMARY:
Dyspnea is common symptom in pulmonary diseases, like chronic obstructive pulmonary disease (COPD) or other pulmonary disease. Ambulatory oxygen therapy is often prescribed to these patients. In these patients resilience, health related quality of life, life satisfaction are measured and the effect and patient satisfaction to ambulatory oxygen therapy are studied.

DETAILED DESCRIPTION:
Dyspnea is a common symptom in pulmonary disease patients, such as chronic obstructive pulmonary disease (COPD) and interstitial lung diseases. These patients often have low health-related quality of life (HRQoL) and life satisfaction (LS), and high levels of anxiety and depression.

Oxygen therapy is used in severe pulmonary diseases to improve HRQoL and prolong survival. Ambulatory oxygen therapy is prescribed to patients who become transiently hypoxemic, e.g. during exercise or normal outdoors activities. However, only 46 % of COPD patients were adherent to long-term oxygen therapy. Proper adaptation to a serious illness, such as advanced COPD and interstitial lung diseases, necessitates resilience. Resilience is an ability to adapt appropriately in difficulties in life. This ability is based on a person's psychological resources, and it can be learned and improved with time and effort. Evaluation of resilience is commonly applied in psychological examinations and research, but less attention has been paid in medical context even though resilience capacity is closely connected to recovery abilities and adaptation.

The main aim is to measure resilience in pulmonary disease patients receiving ambulatory oxygen therapy and how it correlates with other measures of HRQoL and LS. Also anxiety and depression are surveyed and satisfaction to ambulatory oxygen therapy devices and associated services.Investigators also compare the HRQoL of pulmonary disease patients receiving ambulatory oxygen therapy to an age and gender matched sample of the general population. Primary outcome measure was the proportion of patients with low resilience, and secondary outcomes were how resilience correlated with HRQoL, LS, anxiety and depression in patients prescribed ambulatory oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pulmonary disease (e.g. COPD) who has ambulatory oxygen
* Patient with pulmonary disease (e.g. COPD) who is starting to use ambulatory oxygen
* Adult patient
* Informed consent of the patient received

Exclusion Criteria:

* Ambulatory oxygen prescribe for treatment of other than pulmonary disease.
* Age less than 18 years
* Dementia or other cognitive impairment that disables understanding of the study
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary disease who start or use ambulatory oxygen therapy
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Baseline (Before start of ambulatory oxygen therapy)
  15-D - health related quality of life measurement (0= the worst quality of life, 1= the best quality of life)
Health related quality of life | At 24 months
  15-D - health related quality of life measurement (0=the worst quality of life, 1= the best quality of life)

SECONDARY OUTCOMES:
Life satisfaction | Baseline (Before start of ambulatory oxygen therapy)
  Life satisfaction questionnaire (4-6 satisfied, 7-11 partly unsatisfied, 12-20 unsatisfied to life)
Life satisfaction | At 24 months
  Life satisfaction questionnaire (4-6 satisfied, 7-11 partly unsatisfied, 12-20 unsatisfied to life)
Usability of ambulatory oxygen | At one month
  QUEST- questionnaire (The Quebec User Evaluation of Satisfaction with Assistive Technology) (1=unsatisfied, 4-5 very satisfied)
Anxiety | Baseline (Before start of ambulatory oxygen therapy)
  GAD-7 (General Anxiety Disorder-7)- questionnaire (GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety)
Anxiety | 24 months
  GAD-7- questionnaire (General Anxiety Disorder-7) (GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety)
Depression | Baseline (Before start of ambulatory oxygen therapy)
  General Health Questionnaire12 (1= worse or much worse that usually, 0= as usual/much better than usual, points: 0-12, 3 or more points = depression and DEPS- (depression scale) questionnaires (0-30 points, 12 points means that 50% have depression
Depression | At 24 months
  General Health Questionnaire 12 (1= worse or much worse that usually, 0= as usual/much better than usual, points: 0-12, 3 or more points = depression and DEPS- questionnaires (0-30 points, 12 points means that 50% have depression
Sleepiness | Baseline (Before start of ambulatory oxygen therapy)
  Epworth Sleepiness Scale, ESS (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Sleepiness | At 24 months
  Epworth Sleepiness Scale, ESS (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, V, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isokaanta S, Kokki H, Sintonen H, Kokki M. Resilience and health-related quality of life in patients with pulmonary diseases receiving ambulatory oxygen therapy - 24-month follow-up results. BMC Pulm Med. 2025 Jul 4;25(1):326. doi: 10.1186/s12890-025-03778-8. PMID 40616033
- [Derived] Isokaanta S, Honkalampi K, Kokki H, Sintonen H, Kokki M. Resilience and health-related quality of life in patients with pulmonary diseases receiving ambulatory oxygen therapy. BMC Pulm Med. 2021 May 1;21(1):144. doi: 10.1186/s12890-021-01515-5. PMID 33933036